CLINICAL TRIAL: NCT07207720
Title: Respiratory Oscillometry - Establishing Reference Values in Polish Children and Adolescents Aged 3-18 Years (OSCILLONiCA-PL-Kids)
Brief Title: Respiratory Oscillometry Norms for Polish Children and Adolescent.
Acronym: OSCILLONiCA-PL
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Eliza Wasilewska, MD PhD, Medical University of Gdansk
Other Study IDs: OSCILLONiCA-PL-Kids 01/2023
Record Dates: First submitted 2025-09-22; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Healthy; Pulmonary Function Test
Keywords: Reference Values; Oscillometry; Impulse Oscillometry; Respiratory Mechanics; Children; Adolescents; Poland; pulmonary function test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to establish normative values for respiratory oscillometry in the Polish pediatric population. It is designed as a multicentre, population-based, prospective cohort study including children and adolescents aged 3-18 years. The results will provide reference standards for respiratory oscillometry that may support the diagnosis and monitoring of respiratory diseases in clinical practice and research.

DETAILED DESCRIPTION:
OSCILLONiCA-PL-Kids is a multicentre, observational, cross-sectional study designed to establish normative reference values for respiratory oscillometry (IOS) in healthy Polish children and adolescents aged 3-18 years. The study is coordinated by the Polish Society of Pediatric Pulmonology and conducted in 12 pediatric centers across Poland between 2023 and 2025.

Standardized Jaeger oscillometry systems (ERS-validated) are used across all sites, following harmonized operating procedures. All investigators and technicians undergo centralized training and certification, with periodic audits and refresher sessions to ensure procedural consistency and data quality. Measurements are performed during tidal breathing with cheek support and a nose clip, recording at least three technically acceptable trials per participant. Parameters include resistance (Rrs) and reactance (Xrs) at 5, 10, and 20 Hz, resonance frequency (Fres), and area of reactance (AX).

Anthropometric data (height, weight, age, sex) are collected simultaneously to allow modeling of predicted values. Data integrity is verified using automated quality-control algorithms. Reference equations for oscillometric parameters will be derived using generalized additive models for location, scale, and shape (GAMLSS, LMS method). Model performance will be evaluated using the Schwarz Bayesian Criterion, with sensitivity analyses assessing robustness to borderline cases and environmental exposures.

Raw measurement data, as well as derived parameters (means, standard deviations, percentiles, and z-scores), will be used to generate normative reference values and percentile charts stratified by age, height, and sex.

Quality assurance: Data collection and management follow standardized operating procedures (SOPs) approved by the coordinating center. Each site conducts internal data validation prior to upload, and periodic cross-site audits are performed to ensure compliance and consistency. Automatic range and logic checks are implemented in the database to flag out-of-range or inconsistent entries.

Missing data plan: Incomplete or invalid recordings will be excluded from normative modeling. Sensitivity analyses will evaluate the impact of missing data on reference equations. Imputation will not be used for normative dataset derivation.

The study adheres to ERS Technical Standards for Oscillometry (2020) and complies with Good Clinical Practice for observational research. The resulting reference equations and percentile charts will provide validated normative standards for pediatric oscillometry in Poland and support future international harmonization efforts.

ELIGIBILITY:
Inclusion Criteria:1. Age between 3 and 18 years. 2. Caucasian race (Born and residing in Poland). 3. Absence of chronic respiratory disease or acute respiratory symptoms at the time of testing.

4. Written informed consent from a parent/legal guardian (for participants <16 years) or from the participant if ≥16 years.

-

Exclusion Criteria:1. History of chronic lung disease (e.g., asthma, cystic fibrosis, bronchopulmonary dysplasia, interstitial lung disease).

2. Acute respiratory infection within 4 weeks before testing. 3. Severe chronic comorbidities (e.g., congenital heart disease, neuromuscular disorders).

4. Chest deformation 5. Inability to perform oscillometry according to ERS standards.

-

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy Polish children and adolescents aged 3 to 18 years. Participants are recruited from schools, kindergartens, and pediatric outpatient clinics across 12 centers in Poland. Only individuals without chronic respiratory diseases or recent respiratory infections are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Reference values and z-score distributions for respiratory oscillometry parameters (Rrs, Xrs, Fres, AX) in healthy Polish children and adolescents | Single assessment at baseline (during one study visit).
  Quantitative reference data for respiratory oscillometry parameters - respiratory resistance (Rrs) and reactance (Xrs) at 5, 10, and 20 Hz, resonance frequency (Fres), and area of reactance (AX) - measured using impulse oscillometry (IOS) in healthy children and adolescents aged 3-18 years.
  Results will be summarized as mean (Units of Measure:
  Rrs, Xrs: kPa·s·L-¹; Fres: Hz; AX: kPa·L-¹); standard deviation (SD), percentiles, and z-score distributions stratified by age, height, and sex.

SECONDARY OUTCOMES:
Prediction equations and z-score reference models for oscillometric parameters (Rrs, Xrs, Fres, AX) | At baseline (single study visit).
  Regression models describing the relationship between oscillometric parameters (Rrs, Xrs, Fres, AX) and anthropometric predictors (age, height, weight, sex). Models will be developed using the Generalized Additive Models for Location, Scale, and Shape (GAMLSS; LMS method).
  Predicted means, SDs, and z-score equations will be reported, together with model coefficients, standard errors, and model fit indices (Schwarz Bayesian Criterion). Units of Measure: Model coefficients (unitless); Rrs, Xrs: kPa·s·L-¹; Fres: Hz; AX: kPa·L-¹; z-scores: dimensionless
Variability of respiratory oscillometry parameters (Rrs, Xrs, Fres, AX) across pediatric age groups | At baseline (single study visit).
  Mean and standard deviation of oscillometry parameters - respiratory resistance (Rrs, kPa·s·L-¹), reactance (Xrs, kPa·s·L-¹), resonance frequency (Fres, Hz), and area of reactance (AX, kPa·L-¹) - compared across three predefined pediatric age groups: preschool (3-5 years), school-aged (6-12 years), and adolescents (13-18 years).
  All parameters will also be expressed as z-scores (dimensionless) for standardized inter-group comparison.Units of Measure: Rrs, Xrs: kPa·s·L-¹; Fres: Hz; AX: kPa·L-¹; z-scores: dimensionless.
Z-score distributions for oscillometry parameters across Polish and international pediatric cohorts | Up to 24 months after completion of data collection (estimated by December 2026).
  Z-score distributions for respiratory resistance (Rrs), reactance (Xrs), resonance frequency (Fres), and area of reactance (AX) derived from the OSCILLONiCA-KIDS dataset and published international reference datasets (Austria).
  Differences between cohorts will be summarized as mean z-score differences and limits of agreement.
Nomograms and percentile charts for clinical use | Through study completion, approximately 36 months after study start (January 2023 - December 2025).
  Nomograms and percentile charts illustrating predicted oscillometry parameters (Rrs, Xrs, Fres, AX) across age, height, and sex categories will be created to support clinical interpretation. Each chart will include mean, standard deviation (SD), percentiles (5th, 25th, 50th, 75th, 95th), and corresponding z-score ranges.Units of Measure: Rrs, Xrs: kPa·s·L-¹; Fres: Hz; AX: kPa·L-¹; z-scores: dimensionless
De-identified reference dataset of pediatric oscillometry measurements | Through study completion, approximately 36 months after study start (January 2023 - December 2025).
  A de-identified dataset containing oscillometry and anthropometric data (age, height, weight, sex, Rrs, Xrs, Fres, AX) will be compiled for research use and potential integration into international reference initiatives (e.g., Global Lung Function Initiative). Dataset records will be reported as counts of included participants and data completeness metrics. Units of Measure: Number of data records (n); data completeness (%)
Quality and performance indicators of school-based oscillometry testing | Throughout data collection, approximately January 2023 - June 2025.
  Proportion of technically acceptable recordings, coefficient of variation (CoV) between repeated trials, and proportion of children successfully completing valid measurements during school-based testing sessions. Units of Measure:
  Percentage of valid recordings (%); coefficient of variation (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdańsk, Gdansk, Gdańsk, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The study team will consider sharing de-identified individual participant data after publication of the primary results, depending on institutional policies and ethical approval.

REFERENCES:
- [Background] Kaminsky DA, Simpson SJ, Berger KI, Calverley P, de Melo PL, Dandurand R, Dellaca RL, Farah CS, Farre R, Hall GL, Ioan I, Irvin CG, Kaczka DW, King GG, Kurosawa H, Lombardi E, Maksym GN, Marchal F, Oostveen E, Oppenheimer BW, Robinson PD, van den Berge M, Thamrin C. Clinical significance and applications of oscillometry. Eur Respir Rev. 2022 Feb 9;31(163):210208. doi: 10.1183/16000617.0208-2021. Print 2022 Mar 31. PMID 35140105
- [Background] King GG, Bates J, Berger KI, Calverley P, de Melo PL, Dellaca RL, Farre R, Hall GL, Ioan I, Irvin CG, Kaczka DW, Kaminsky DA, Kurosawa H, Lombardi E, Maksym GN, Marchal F, Oppenheimer BW, Simpson SJ, Thamrin C, van den Berge M, Oostveen E. Technical standards for respiratory oscillometry. Eur Respir J. 2020 Feb 27;55(2):1900753. doi: 10.1183/13993003.00753-2019. Print 2020 Feb. PMID 31772002
- [Background] Desai U, Joshi JM. Impulse oscillometry. Adv Respir Med. 2019;87(4):235-238. doi: 10.5603/ARM.a2019.0039. PMID 31476011
- [Background] de Oliveira Jorge PP, de Lima JHP, Chong E Silva DC, Medeiros D, Sole D, Wandalsen GF. Impulse oscillometry in the assessment of children's lung function. Allergol Immunopathol (Madr). 2019 May-Jun;47(3):295-302. doi: 10.1016/j.aller.2018.03.003. Epub 2018 Jul 5. PMID 29983239
- See also: This external link directs to the official website of the Polish Society of Pediatric Pulmonology (PTPD), which provides information about the OSCILLONiCA-PL Kids study. The page contains a public description of the project "Respiratory Oscillometry - Es — https://ptpd.edu.pl/nowe-wpisy/oscylometria-ukladu-oddechowego-opracowanie-norm-populacyjnych-dla-dzieci-i-mlodziezy-w-wieku-3-18-lat/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT07207720/Prot_SAP_ICF_000.pdf